CLINICAL TRIAL: NCT02516579
Title: ESCORT-HU : European Sickle Cell Disease Cohort - Hydroxyurea
Brief Title: European Sickle Cell Disease Cohort - Hydroxyurea
Acronym: ESCORT-HU
Status: Completed | Type: Observational
Sponsor: Theravia (Industry)
Responsible Party: Sponsor
Other Study IDs: ESCORT-HU
Record Dates: First submitted 2015-07-23; First posted 2015-08-06 (Estimated); Results first posted 2020-03-19 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Siklos
  Other Names: hydrocarbamide

SUMMARY:
In the context of the Risk Management Plan (RMP), as requested from Addmedica by the EMEA, to collect information about long-term safety of Siklos® (hydroxycarbamide) when used in patients with Sickle Cell Disease.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ambulatory patients, aged 2 years and more (children, adolescents or adults)
* With symptomatic sickle cell syndrome
* Treated with Siklos®
* Having been informed of the study by the initiating physician and consenting to participate to the cohort.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient with sickle-cell disease
Sampling Method: Non-Probability Sample
Enrollment: 1906 (Actual)
Dates: Start 2009-01; Primary Completion 2019-03-20 (Actual); Study Completion 2019-03-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Galacteros, MD, Principal Investigator — Hôpital henri Mondor (Adults); Mariane de Montalembert, MD, Principal Investigator — Hôpital Necker Enfants Malades (Children)
Locations (60):
- France (41):
  - CHU d'Amiens - Picardie - Site sud, Amiens
  - Centre Hospitalier Robert Ballanger, pédiatrie et néonatalogie, Aulnay-sous-Bois
  - Hôpital Avicenne; médecine interne, Bobigny
  - Hôpital Jean Verdier; médecine interne, Bondy
  - Hôpital Jean Verdier; pédiatrie, Bondy
  - CHU Bordeaux, urgences pédiatriques, Bordeaux
  - Hôpital Saint-André, Bordeaux
  - CHU Estaing, pédiatrie, Clermont-Ferrand
  - Hôpital Louis Mourier; pédiatrie, Colombes
  - Hôpital Louis Mourier; service de pédiatrie, Colombes
  - Centre hospitalier intercommunal de Créteil, Créteil
  - Hôpital Henri Mondor, centre de la Drépanocytose, Créteil
  - Centre Hospitalier de Gonesse, médecine interne, Gonesse
  - Centre Hospitalier de Gonesse, pédiatrie, Gonesse
  - CHU de Grenoble, hôpital Couple Enfant, Grenoble
  - CHU de Grenoble, Grenoble
  - CHU de Limoges, Limoges
  - Hôpital Mère-Enfant, Limoges
  - Hôpital Edouard Herriot, hémovigilance, Lyon
  - Institut d'Hématologie et d'Oncologie Pédiatrique, Lyon
  - CHU Timone, Marseille
  - Hôpital de la Conception, médecine interne, Marseille
  - Centre Hospitalier Intercommunal André Grégoire, Montreuil
  - CHU Nantes, Hôpital Hôtel Dieu, Nantes
  - Hôpital Trousseau; pédiatrie générale, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - Hôpital Necker enfants, maladies infectieuses et tropicales, Paris
  - Hôpital Necker; biothérapie, Paris
  - Hôpital Necker; maladies infectieuses et tropicales, Paris
  - Hôpital Robert Debré, immunologie-hématologie pédiatrique, Paris
  - CHR Reims, American Memorial Hospital, Reims
  - CHU Rennes, Hôpital Pontchaillou, Rennes
  - CHU Rennes, hôpital Sud, Rennes
  - CHU Charles Nicolle, Rouen
  - CHU de Rouen - Hôpital Charles Nicolle, Rouen
  - Centre Hospitalier Delafontaine, médecine interne, Saint-Denis
  - Centre Hospitalier Delafontaine, pédiatrie, Saint-Denis
  - CHRU Strasbourg, Hôpital de Hautepierre, Strasbourg
  - CHU Toulouse; hôpital des enfants, Toulouse
  - Institut Universitaire du cancer; médecine interne, Toulouse
  - CHU Nancy, Brabois enfants, Vandœuvre-lès-Nancy
- French Guiana (3):
  - CH André Rosemon, Cayenne
  - CMCK, Kourou
  - CH Ouest Guyanais, Saint-Laurent-du-Maroni
- Germany (6):
  - Charité-Universitätsmedizin, Berlin, Berlin
  - Pädiatrie Klinikum Delmenhorst, Delmenhorst
  - Heinrich-Heine Universität Düsseldorf, Düsseldorf
  - University of Freiburg, Freiburg im Breisgau
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - München, München
- Laiko General Hospital, Athens, Greece
- Guadeloupe (3):
  - CH Basse-Terre, adultes, Basse-Terre
  - CH Basse-Terre, enfants, Basse-Terre
  - CHU Pointe à Pitre, Pointe-à-Pitre
- Italy (3):
  - Clinica Pediatrica AOU, Napoli
  - Azienda Ospedaliera-University of Padova, Padua
  - Azienda Ospedaliera Universitaria Integrata (AOUI Verona), Verona
- Martinique (3):
  - CHU Fort de France, Fort-de-France
  - Hôpital Pierre Zobda-Quitman, Fort-de-France
  - CH Lamentin, Le Lamentin

REFERENCES:
- [Derived] Allali S, Galacteros F, Oevermann L, Cannas G, Joseph L, Loko G, Elenga N, Benkerrou M, Etienne-Julan M, Castex MP, Brousse V, de Montalembert M. Hydroxyurea is associated with later onset of acute splenic sequestration crisis in sickle cell disease: Lessons from the European Sickle Cell Disease Cohort-Hydroxyurea (ESCORT-HU) study. Am J Hematol. 2024 Apr;99(4):555-561. doi: 10.1002/ajh.27214. Epub 2024 Jan 22. PMID 38247384
- [Derived] de Montalembert M, Voskaridou E, Oevermann L, Cannas G, Habibi A, Loko G, Joseph L, Colombatti R, Bartolucci P, Brousse V, Galacteros F; All ESCORT HU Investigators. Real-Life experience with hydroxyurea in patients with sickle cell disease: Results from the prospective ESCORT-HU cohort study. Am J Hematol. 2021 Oct 1;96(10):1223-1231. doi: 10.1002/ajh.26286. Epub 2021 Jul 23. PMID 34224583

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients With Sickle Cell Disease Treated With Siklos®: The follow-up of the patients was strictly observational and fitted within their usual clinical monitoring without any controlled treatment, specific exam or modification of their follow-up, in compliance with the Summary of Product Characteristics of the product.
Period: Overall Study
Arm/Group | Patients With Sickle Cell Disease Treated With Siklos®
Started | 1906
Completed | 1906
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 1906 patients included but 1903 patient took at least one dose of Siklos and are included in the analysis
Arm/Group | Patients With Sickle Cell Disease Treated With Siklos®
Number analyzed (Participants) | 1903
Age, Continuous [Median (Full Range); unit: years] — Population: 1906 patients were included but 1903 patients took at least one dose of Siklos and were included in the analysis
  years | 21.4 [0.8 to 70.4]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 1906 patients were included but 1903 patient took at least one dose of Siklos and were included in the analysis
  Participants
    Female | 1051
    Male | 852
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants] — Population: 1906 patients were included but 1903 took at least one dose of Siklos and were included in the analysis
  participants
    Greece | 173
    Italy | 10
    France | 1575
    Germany | 145

OUTCOME MEASURES:

1. Primary Outcome: % of Patient-years With Malignancies
Time Frame: During the follow-up of participant, up to 10 years
Population: Patients with follow-up visit
Measure: Number; unit: % patient-years
Arm/Group | Patients With Sickle Cell Disease Treated With Siklos®
Number analyzed (Participants) | 1854
% patient-years | 0.001

2. Primary Outcome: % of Patient-years With Skin Ulcerations
Description: Patients with at least one skin ulceration
Time Frame: During the follow-up of participant, up to 10 years
Measure: Number; unit: % patient-years
Arm/Group | Patients With Sickle Cell Disease Treated With Siklos®
Number analyzed (Participants) | 1854
% patient-years | 1.13

3. Primary Outcome: % of Patient-years With Myelosuppressions
Description: Patients with at least one myelosuppression
Time Frame: During the follow-up of participant, up to 10 years
Measure: Number; unit: % patient-years
Arm/Group | Patients With Sickle Cell Disease Treated With Siklos®
Number analyzed (Participants) | 1854
% patient-years | 5.99

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the follow-up of participant, up to 10 years
Arm/Group | Patients With Sickle Cell Disease Treated With Siklos®
All-Cause Mortality (participants affected / at risk) | 33/1903
Serious Adverse Events (participants affected / at risk) | 705/1903
Other Adverse Events (participants affected / at risk) | 1308/1903
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patients With Sickle Cell Disease Treated With Siklos® (N=1903)
infections and infestations (Infections and infestations) | 346
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 155
respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 151
general disorders and administration site conditions (General disorders) | 97
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patients With Sickle Cell Disease Treated With Siklos® (N=1903)
infections and infestations (Infections and infestations) | 645
General disorders and administration site conditions (General disorders) | 386
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 370

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-20): https://cdn.clinicaltrials.gov/large-docs/79/NCT02516579/Prot_SAP_000.pdf